CLINICAL TRIAL: NCT03100110
Title: NeuroCognitive Communicator Exploratory Safety Study of an Assistive Neuroprosthetic Device for Patients With Severe Upper Motor Disability.
Brief Title: NeuroCognitive Communicator: Safety Study
Acronym: NCC-1701
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 20170100-01H
Record Dates: First submitted 2017-02-21; First posted 2017-04-04 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Motor Neuron Disease, Amyotrophic Lateral Sclerosis; Tetraplegia
Keywords: Brain-Computer Interface; Brain-Machine Interface; Prefrontal Cortex
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Quadriplegia | interventions — Brain-Computer Interfaces

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NeuroCognitive Communicator (Experimental)
  Interventions: Device: NeuroCognitive Communicator

INTERVENTIONS:
Device: NeuroCognitive Communicator — Comprises an electrode array in prefrontal cortex, another in motor cortex, Blackrock NeuroPort system and connectors, augmentative assistive communication application, robotic arm, and virtual reality environment.
  Other Names: Utah Array; Blackrock Microsystems NeuroPort; Brain-Computer Interface; Brain-Machine Interface

SUMMARY:
Individuals suffering from tetraplegia as a result of cervical spinal cord injury, brainstem stroke, or amyotrophic lateral sclerosis (ALS) cannot independently perform tasks of daily living. In many cases, these conditions do not have effective therapies and the only intervention is the provision of assistive devices to increase independence and quality of life. However, currently available devices suffer from usability issues and are limiting for both the patient and caregiver. One of the most progressive alternative strategies for assistive devices is the use of brain-computer interface (BCI) technology to translate intention signals directly from sensors in the brain into computer or device action. Preclinical primate research and recent human clinical pilot studies have demonstrated success in restoring function to disabled individuals using sensors implanted directly in motor regions of the brain. Other preclinical primate research has demonstrated effective intention translation from sensors implemented in cognitive regions of the brain and that this information complements information from the motor regions. The current proposal seeks to build on these studies and to test the safety aspects related to implanting two sensors, each a microelectrode array, into both the motor and cognitive regions of the brain in motor impaired humans. Secondary objectives include feasibility evaluation of the complementary sensors in their ability to support effective assistive communication.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of a complete or incomplete cervical spinal cord injury, with stable neurological deficits greater than 1 year, or ALS with equivalent degree of deficit.
* Maintain some level of communication, enough to independently provide informed consent for the study.
* Deemed healthy for surgery.
* Good psychological and social stability.
* Prospective participants with ALS must already have an advanced directive with regard to ventilation.
* Live within a one-hour travel duration of the site.

Exclusion Criteria:

* Presence of previous certain implanted devices.
* In the opinion of the investigator, the presence of other serious disease or disorder that could affect ability to participate in this study.
* Ongoing participation in another clinical trial.
* Individuals who are immunosuppressed or who have conditions that typically result in immunocompromise (eg. chronic corticosteroid use, immunomodulators, chemotherapy).
* Presence of clinical depression that is not medically optimized, as screened by a neuropsychologist on our team.
* Presence of cognitive deficits, as assessed by a neuropsychologist on our team, that would preclude completion of some cognitively challenging tasks.
* The participant has plans to move outside the study radius within the study period.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2019-05-13 (Actual); Primary Completion 2024-04-15 (Estimated); Study Completion 2024-04-15 (Estimated)

PRIMARY OUTCOMES:
Rate of adverse events | 6 months
  Transcutaneous connector will be assessed by physician 3-4 times per week for skull and scalp health and lack of infection.
  All adverse events associated with the system will be measured.
Change in quality of life as assessed by McGill Quality of Life questionnaire. | 6 months
  McGill Quality of Life questionnaire will be administered monthly; shortened version will be administered 3-4 times per week.

SECONDARY OUTCOMES:
Percentage of allotted time spent with each augmentative and assistive communication technology. | 6 months
  At the end of most experimental sessions, the participant will have time to operate the NCC to control augmentative and assistive communication (AAC) technologies such as robotic arms or spellers. We will measure the percentage of allotted time that the participant spends operating each AAC technology, or choosing not to operate any AAC technology. The data will be aggregated across all AAC sessions with time allotted to AAC operation.
Information transfer rate (measured in bits per second) achieved by each participant calculated during closed-loop operation of the neuroprosthetic device, aggregated across trials within a task. | 6 months
  Participants will perform repeated trials of experimental tasks designed to activate recorded brain regions. Task progression will be modulated by neuronal activity. Successful completion of the task will require volitional modulation of neuronal activity. Task performance will be quantified by the information transfer rate which is calculated from the number of bits of information communicated by each trial's selection(s) and the amount of time it took to complete a trial.
Coefficients of neuronal activity covariance matrix and their dependence on task performance. | 6 months
  Neuronal activity time series covary across neurons within a brain region and across brain regions. The degree of covariance will be recorded in the coefficients of the covariance matrix, scaled from -1 to +1. The covariance matrix will be recorded under different task conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No